CLINICAL TRIAL: NCT00692354
Title: A Phase I Study to Evaluate the Safety and Tolerability, of the Aminopeptidase Inhibitor, CHR-2797, in Patients With Advanced Tumours
Brief Title: Safety Study to Evaluate CHR-2797 in Patients With Advanced Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chroma Therapeutics (Industry)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Dr Leon Hooftman, Chroma Therapeutics Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-2797-001
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2008-06

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced; Solid; Tumour; Tumor; Oral
MeSH Terms: conditions — Neoplasms | interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CHR-2797 (tosedostat) — Drug was given orally, once daily, ensuring a dosing interval of approximately 24 hours. Dose escalations took place starting at 10mg and escalating (per protocol) as follows: 20, 40, 90, 130, 180, 240 and 320 mg

SUMMARY:
The primary objective of this study was to determine the safety, tolerability, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of CHR-2797 when administered orally, once daily, to patients with advanced solid tumours.

The secondary objectives of this study were:

* To determine pharmacokinetic parameters for CHR-2797 when administered orally at increasing dose levels;
* To investigate the pharmacodynamic effects of CHR-2797 in blood mononuclear cells and, when possible, tumour cells; - To enable a preliminary assessment of anti-tumour activity of CHR-2797.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent
* Histological or cytologically confirmed malignant solid tumour refractory to standard therapy or for which no standard therapy exists
* Evaluable disease
* Recovered from the acute adverse effects of prior therapies (excluding alopecia and grade 1 neuropathy)
* Adequate bone marrow, hepatic and renal function including the following:

  1. Hb ≥ 9.0 g/dl, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 100x109/L
  2. Total bilirubin ≤ 1.5 x upper normal limit
  3. AST and ALT ≤ 2.5 x upper normal limit (or ≤ 5 x UNL in the presence of liver metastases)
  4. Creatinine ≤1.5 x upper normal limit
* Age < 18 years
* Performance status (PS) < 2 (ECOG scale)
* Estimated life expectancy greater than 3 months
* Female patients with reproductive potential had to have a negative serum pregnancy test within 7 days of treatment. Both women and men had to agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment. Acceptable methods of contraception included IUD, oral contraceptive, sub-dermal implant and double barrier (condom with a contraceptive sponge or contraceptive pessary)

Exclusion Criteria:

* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 4 weeks prior to study entry (or a longer period depending on the defined characteristics of the agents used e.g. 6 weeks for mitomycin or nitrosourea). In patients with progressive disease (PD), continuation of LHRH agonists for prostate cancer, bisphosphonates for bone disease and corticosteroids was permitted provided the dose was stable before and during the study
* Co-existing active infection or serious concurrent illness
* Significant cardiovascular disease as defined by

  1. History of congestive heart failure requiring therapy
  2. History of unstable angina pectoris or myocardial infarction up to 6 months prior to study entry
  3. Presence of severe valvular heart disease
  4. Presence of a ventricular arrhythmia requiring treatment
* Any co-existing medical condition that in the Investigator's judgement substantially increased the risk associated with the patient's participation in the study
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
* Gastrointestinal disorders that might have interfered with absorption of the study drug
* Persistent grade 2 or greater toxicities from any cause
* Patients with known brain tumours or metastases should have been excluded from this clinical study because of their poor prognosis and because they often develop progressive neurologic dysfunction that would have confounded the evaluation of neurologic and other AEs
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-10; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of CHR-2797 when administered orally, once daily, to patients with advanced solid tumours. | 3 years

SECONDARY OUTCOMES:
To determine the PK parameters for oral CHR-2797 at increasing dose levels; | 3 years
To investigate the PD effects of CHR-2797 in blood and tumour cells | 3 years
To enable a preliminary assessment of anti-tumour activity of CHR-2797 | 3 years